CLINICAL TRIAL: NCT06946680
Title: Phase I Study -To Assess Safety and Feasibility of IL-8 Receptor Modified Patient-derived Activated CD70 CAR T Cell Therapy in CD70+ Adult GBM and Pediatric High-Grade Gliomas (pHGG)
Brief Title: IL-8 Receptor-modified CD70 CAR T Cell Therapy in CD70+ Pediatric High-grade Glioma (HGG)
Acronym: IMPACT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Florida Department of Health, Live Like Bella (Unknown); St. Baldrick's Foundation (Other); American Brain Tumor Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202200057-P; OCR41673 (Other: University of Florida)
Record Dates: First submitted 2025-04-11; First posted 2025-04-27 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: High-grade Glioma
Keywords: CAR T Cell; Brain Tumor; Brain Cancer; Immunotherapy; Glioblastoma
MeSH Terms: conditions — Glioma; Brain Neoplasms; Glioblastoma | interventions — Receptors, Interleukin-8B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 8R-70CAR T cells (Experimental): Cohort 1 will receive 1 x 10^6 cells/kg. Cohort 2 will receive 1 x 10^7 cells/kg. Cohort 3 will receive 1 x 10^8 cells/kg.
  Interventions: Biological: Ex-Vivo expanded autologous IL-8 receptor (CXCR2) modified CD70 CAR (8R-70CAR) T cells

INTERVENTIONS:
Biological: Ex-Vivo expanded autologous IL-8 receptor (CXCR2) modified CD70 CAR (8R-70CAR) T cells — Single dose of 8R-70CAR T cells administered IV
  Other Names: 8R-70CAR T cells

SUMMARY:
This is a phase I study to assess the safety and feasibility of IL-8 receptor modified patient-derived activated CD70 CAR T cell therapy in CD70+ pediatric high-grade glioma

DETAILED DESCRIPTION:
Identified newly-diagnosed pediatric CD70+ HGG patients will be enrolled in this clinical trial study prior to initiation of standard-of-care chemo-radiation. Prior to initiation of chemoradiation, PBMCs will be collected through peripheral venipuncture. After tumor CD70 status is confirmed, the 8R-70CAR T cell production will start.

4 weeks (+/- 1) post completion of radiation, pediatric patients, based on institutional policy, will initiate adjuvant chemo with dose-intensified TMZ 75-100 mg/m2/day x 21 days for up to 3 cycles. 8R-70CAR T cells will be administered at day 21-24 of the TMZ cycle as a single intravenous (IV) infusion, or for pediatric patients not receiving adjuvant chemo once 8R-70CAR T cells. Pediatric patients will receive lymphodepletion prior to CAR T cell administration.

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed pHGG based on the absence of a previous history of brain tumor (WHO Grade III-IV glioma) by histopathology.
* CD70 positive (≥5%, 1+) The tumors from the surgical resection or biopsy by immunohistochemistry will be confirmed by a validated assay performed at UF Health Pathology, a certified Lab.

  o CD70 tumor expression performed on paraffin-embedded tumor specimens will be evaluated. Tumor expression will be scored on a scale of 0 to 3 staining intensity: 0 = Negative
  1. = Low level
  2. = Moderate level
  3. = High level The criteria for inclusion will be at least 5% of the cells scoring 1+ staining intensity (> 5%, 1+).
* Karnofsky Performance Status (KPS) or Lansky Performance Score (LPS) of > 70% Patients who are unable to walk because of neurologic deficits, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score provided the neurological deficit is stable.
* CBC with differential with adequate bone marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1000 cells/mm3.
  * Platelet count ≥ 100,000 cells/mm3.
  * Hemoglobin ≥ 10 g/dl. (The use of transfusion or other intervention to achieve Hgb ≥ 10 g/dl is acceptable.)
* Adequate renal function as defined below:

  o Serum creatinine < 1.5 x institutional upper limit of normal for age and gender. Patients who do not meet the criteria but have a 24-hour Creatinine Clearance or GFR (radioisotope or iothalamate) ≥ 70 mL/min/1.73 m2 are eligible
* Adequate hepatic function as defined below:

  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) for age
  * ALT ≤ 3 times institutional upper limits of normal for age
  * AST ≤ 3 times institutional upper limits of normal for age
* Signed informed consent, or for patients age <18, parental permission, and, as appropriate, assent from pediatric patients age ≥12. If the patient's mental status precludes their informed consent, the legally authorized representative may give informed consent. Consent or permission/assent will be obtained at screening (before PBMC collection) and before treatment with CAR T-cells.
* For females of childbearing potential, a negative serum pregnancy test at enrollment.
* Women of childbearing potential (WOCBP) must be willing to use an acceptable contraceptive method to avoid pregnancy throughout the study and for at least 24 weeks after the last dose of study drug.
* Males with female partners of childbearing potential must agree to practice adequate contraceptive methods throughout the study and should avoid conceiving children for 24 weeks following the last dose of study drug.

Exclusion Criteria:

* Prior invasive malignancy (except for non-melanomatous skin cancer) unless disease free for ≥ 3years. (In situ cancer is permissible)
* Spinal metastasis and leptomeningeal involvement.
* Patients with Bulky Tumors:

  * 3 cm in a single dimension (post-surgery)
  * Tumor causing uncal herniation or mass effect leading to midline shift with or without symptoms or signs of impending herniation or
  * Obstruction to CSF flow
* Recurrent or multifocal malignant gliomas.
* The patient is not a candidate for cellular therapy as assessed by the study bone marrow transplant physician.
* Known immunosuppressive disease or human immunodeficiency virus (HIV) infection.

HIV-positive patients are ineligible due to the unknown safety and efficacy of infusing these patients with CAR T cells genetically modified using retroviral vectors. Additionally, the immunosuppression used for treatment in this study will pose an unacceptable risk.

• Concurrent illness: Patients with active autoimmune disease, documented history of autoimmune disease/syndrome, or any other condition that requires ongoing systemic steroids or systemic immunosuppressive agents, except

* Patients with vitiligo or resolved asthma/atopy
* Patients with hypothyroidism stable on hormone replacement or Sjogren's syndrome
* Patients requiring physiologic doses of corticosteroids (up to 0.5 mg/m2/day dexamethasone equivalent)

  * History of or ongoing pneumonitis or significant interstitial lung disease.
  * Ongoing or active uncontrolled infection.
  * Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the opinion of the investigator, would compromise the patient's ability to tolerate protocol therapy, put them at additional risk for toxicity or would interfere with the study procedures or results.
  * Patients with any of the following cardiac diseases:
* New York Heart Association (NYHA) functional class III or IV
* Clinically significant cardiac arrhythmia including, but not limited to, Torsade de pointes or requiring a pacemaker
* Left ventricular ejection fraction below 50% as determined by echocardiography (ECHO)

  * Pregnant or lactating women, due to possible adverse effects on the developing fetus or infant.
  * Patients treated on any other therapeutic clinical protocols within 30 days prior to enrollment.
  * For females of childbearing potential, a negative serum pregnancy test at enrollment.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2045-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of investigational treatment related severe toxicity (Dose-limiting toxicity event) | administration of 8R-70CAR T to 28 days post-infusion
  Safety is defined as the adverse events (AEs), serious adverse events (SAEs) and dose-limiting toxicities (DLT) observed throughout the trial.
Prevalence of enrolled subjects who receive a qualified immunotherapy investigational product. | Enrollment up to 18 weeks
  Feasibility will be measured by the number of patients who receive 8R-70CAR T-cell that met the FDA IND defined quality assurance and quality control release criteria. A minimum of 66.7 % of enrolled subjects must achieve this criterion for the feasibility endpoint.
Maximum tolerated dose (MTD) dose-finding endpoint based on Dose-Limiting-Toxicity (DLT) incidence | administration of 8R-70CAR T to 28 days post-infusion
  Determination of the maximum tolerated dose (MTD) of 8R-70CAR T cells based on the incidence of investigational treatment-related severe toxicity (dose-limiting toxicity events)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Ghiaseddin, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Health Children's Hospital, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No